CLINICAL TRIAL: NCT00103779
Title: A Phase I, Multi-Dose Study of SGN-40 (Anti-huCD40 mAb) in Patients With Non-Hodgkin's Lymphoma
Brief Title: A Safety Study of SGN-40 in Patients With Non-Hodgkin's Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Seagen Inc. (Industry)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Jonathan Drachman, MD, Seattle Genetics, Inc.
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SG040-0002
Expanded Access: Available
Record Dates: First submitted 2005-02-14; First posted 2005-02-15 (Estimated); Last update posted 2014-12-18 (Estimated); Status verified 2014-12

CONDITIONS: Non-Hodgkin Lymphoma
Keywords: Antigens, CD40; Antibody, Monoclonal; Lymphoma, Non-Hodgkin; Lymphoma, B-Cell; Hematologic Diseases; Immunoproliferative Disorders; Lymphatic Diseases; Lymphoproliferative Disorders; Lymphoma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Lymphoma, B-Cell; Hematologic Diseases; Immunoproliferative Disorders; Lymphatic Diseases; Lymphoproliferative Disorders; Lymphoma | interventions — dacetuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: SGN-40 (anti-huCD40 mAb)

INTERVENTIONS:
Drug: SGN-40 (anti-huCD40 mAb) — 1 mg/kg IV (in the vein) on Day 1; 1-2 mg/kg IV on Day 4; 2-4 mg/kg IV on Day 8; 3-8 mg/kg on Days 15, 22 and 29.
  Other Names: dacetuzumab

SUMMARY:
This is an open-label, multi-dose, Phase I, dose escalation study to define the safety profile and preliminary anti-tumor activity of SGN-40 in patients with refractory or recurrent non-Hodgkin B-cell lymphomas.

DETAILED DESCRIPTION:
A minimum of 3 patients will be entered into each dose-level cohort for 5 weeks. A dose-escalation schema will be employed in cohorts. The initial dose starts at 1 mg/kg on Day 1 and 4 followed by 2mg/kg on Day 8. Dose escalation will occur on weeks 3-5 with a maximum weekly dose of 8 mg/kg. Patients who meet criteria of at least partial response will be eligible for additional 4 weekly doses at highest dose tolerated.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a histological diagnosis of B cell non-Hodgkin's lymphoma, including diffuse large B-cell, mantle cell, follicular, small lymphocytic, and marginal zone lymphoma by the World Health Organization criteria.
* Patients must have an archived paraffin or fresh tumor specimen available for immunohistologic evaluation of CD40, CD20, & CD79a.
* Patients must have relapsed lymphoma and must have failed frontline chemotherapy.
* Patients who have not received autologous stem cell transplant must have refused or be ineligible for it.
* Patients must have completed radiotherapy, chemotherapy, and/or treatment with investigational anti-cancer agents 4 weeks prior to registration. Patients must have completed any monoclonal antibody treatment, including rituximab, 6 months prior to registration.
* Patients must have completed autologous bone marrow transplant 4 months prior to registration.
* Patient must have at least one site of measurable disease defined by unidimensional lesion ≥ 2 cm by conventional CT scan.
* Patients must have an ECOG performance status ≤ 2 and a life expectancy > 3 months.
* Patients must have the following required baseline laboratory data:

  * Platelet count ≥ 75,000/mm3,
  * Hemoglobin ≥ 9.0 g/dL,
  * Absolute neutrophil count ≥ 1,250/mm3,
  * ALT/AST ≤ 2.5 times ULN,
  * Total bilirubin ≤ 1.5 times ULN,
  * Creatinine < 1.5 mg/dL,
* Females of childbearing potential must have a negative serum β-hCG pregnancy test result within 3 days prior to the first dose of SGN-40 and must agree to use an effective contraceptive method during the course of the study and for 6 months following the last dose of study drug.
* If a deep venous thrombosis or other vascular even has required medical or surgical intervention in the past year, patients must either be on stable dose of anticoagulant therapy for at least 3 weeks or have completed anticoagulant therapy at least 3 months prior to registration with radiographic confirmation that thrombosis is resolved.
* Patients must be at least 18 years of age.
* Patients must be available for periodic blood sampling, study-related assessments and management of toxicity at the treating institution.

Exclusion Criteria:

* Patients with history or clinical evidence of leptomeningeal or central nervous system (CNS) lymphoma.
* Patients with a documented history within 6 months of registration of a cerebral vascular event, myocardial infarction, deep venous thrombosis or other vascular event that has required medical or surgical intervention. Patients must have completed anticoagulant therapy at least 3 months prior to registration. Prophylactic anticoagulant therapy for indwelling catheters is acceptable.
* Patients who have received an allogeneic stem cell transplant.
* Patients who have had major surgery within 4 weeks prior to registration.
* Patients with a known hypersensitivity to recombinant proteins or any excipient contained in the drug formulation.
* Patients with a history of another primary malignancy that has not been in remission for at least 5 years (non-melanoma skin cancer and cervical carcinoma in situ on biopsy or a squamous intraepithelial lesion on PAP smear are exempt from the five year limit).
* Patients with any active systemic viral, bacterial, or fungal infection within four weeks prior to registration.
* Patients with known positivity for HIV, hepatitis B or hepatitis C infection.
* Patients with a history of significant chronic or recurrent infections requiring treatment.
* Patients with a history of migraines or severe headaches requiring medical therapy within 12 months of enrollment.
* Patients on systemic steroids who have not been on a stable daily dose (not exceeding 10 mg prednisone or equivalent) during 4 weeks prior to the first dose of SGN 40.
* Patients who are pregnant or breastfeeding.
* Patients with any serious underlying medical condition that would impair their ability to receive or tolerate the planned treatment.
* Patients with dementia or altered mental status that would preclude the understanding and/or rendering of informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2004-12; Primary Completion 2007-03 (Actual); Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Adverse events and lab abnormalities.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Drachman, MD, Study Director — Seagen Inc.
Locations (5):
- United States (5):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Stanford University, Stanford, California
  - University of Miami, Miami, Florida
  - Cornell University, New York, New York
  - University of Texas MD Anderson Cancer Center, Houston, Texas

REFERENCES:
- [Result] Advani R, Forero-Torres A, Furman RR, Rosenblatt JD, Younes A, Ren H, Harrop K, Whiting N, Drachman JG. Phase I study of the humanized anti-CD40 monoclonal antibody dacetuzumab in refractory or recurrent non-Hodgkin's lymphoma. J Clin Oncol. 2009 Sep 10;27(26):4371-7. doi: 10.1200/JCO.2008.21.3017. Epub 2009 Jul 27. PMID 19636010
- See also: Related Info — http://www.ncbi.nlm.nih.gov/pubmed/19636010